CLINICAL TRIAL: NCT01977755
Title: A Randomised, Double-Blind, Placebo-Controlled, Parallel-Group Trial to Assess Clinical Efficacy and Safety of Danegaptide in Patients With ST-Elevation Myocardial Infarction Undergoing Primary Percutaneous Coronary Intervention
Brief Title: Phase 2 Clinical Proof-of-Concept Study of the Cardioprotective Properties of Danegaptide in ST Segment Elevation Myocardial Infarction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Zealand Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 13-031
Record Dates: First submitted 2013-10-30; First posted 2013-11-07 (Estimated); Last update posted 2018-04-06 (Actual); Status verified 2016-01

CONDITIONS: Focus of Study is STEMI
MeSH Terms: interventions — danegaptide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- danegapetide high dose (Active Comparator): 7,5 mg bolus injection, followed by 22,5 mg infused over 6 hours
  Interventions: Drug: danegaptide
- danegaptide low dose (Active Comparator): 2,5 mg bolus injection, followed by 7,5 mg infused over 6 hours
  Interventions: Drug: danegaptide
- Placebo (Placebo Comparator): bolus injection, followed by infused over 6 hours
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: danegaptide
  Arms: danegapetide high dose; danegaptide low dose
Drug: Placebo
  Arms: Placebo

SUMMARY:
This study explores the potential cardioprotective properties of danegaptide when administered to patients with ST-Segment elevation myocardial infarction.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* ST-segment elevation myocardial infarction
* Acute onset of chest pain of < 12 hours duration

Exclusion Criteria:

* Pregnancy
* Known prior Myocardial Infarction in same area as present STEMI, known hypertrophic or dilated cardiomyopathy, or prior hospital admission for heart failure
* Contraindication for cardiac MRI
* Inability to understand information or provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 591 (Actual)
Dates: Start 2013-11; Primary Completion 2015-12-20 (Actual); Study Completion 2016-06-08 (Actual)

PRIMARY OUTCOMES:
Myocardial Salvage Index | 3 months
  Myocardial Salvage Index as assessed by MRI and calculated as the difference between myocardial volume at risk and final infarct size in relation to myocardial volume at risk

SECONDARY OUTCOMES:
Relative Infarct size, Absolute Infarct size, Left Ventricular Ejection Fraction (LVEF), microvascular obstruction and infarct haemorrhage as determined by MRI | 3 months
Degree of ST-resolution and fraction of patients with 70 % ST-resolution measured by ECG 60 minutes post Percutaneous Coronary Intervention procedure | 60 minutes
Major Clinical Adverse Events including cardiac death, new or worsening heart failure and re-admission for heart failure | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Engstrom, MD, DMSci, Principal Investigator — The Heart Center, Rigshopitalet University of Copenhagen
Locations (1):
- The Heart Center, Rigshospitalet, University of Copenhagen, Copenhagen, Denmark

REFERENCES:
- [Derived] Thomsen AF, Bertelsen L, Jons C, Jabbari R, Lonborg J, Kyhl K, Goransson C, Nepper-Christensen L, Atharovski K, Ekstrom K, Tilsted HH, Pedersen F, Kober L, Engstrom T, Vejlstrup N, Jacobsen PK. Scar border zone mass and presence of border zone channels assessed with cardiac magnetic resonance imaging are associated with ventricular arrhythmia in patients with ST-segment elevation myocardial infarction. Europace. 2023 Mar 30;25(3):978-988. doi: 10.1093/europace/euac256. PMID 36576342
- [Derived] Engstrom T, Nepper-Christensen L, Helqvist S, Klovgaard L, Holmvang L, Jorgensen E, Pedersen F, Saunamaki K, Tilsted HH, Steensberg A, Fabricius S, Mouritzen U, Vejlstrup N, Ahtarovski KA, Goransson C, Bertelsen L, Kyhl K, Olivecrona G, Kelbaek H, Lassen JF, Kober L, Lonborg J. Danegaptide for primary percutaneous coronary intervention in acute myocardial infarction patients: a phase 2 randomised clinical trial. Heart. 2018 Oct;104(19):1593-1599. doi: 10.1136/heartjnl-2017-312774. Epub 2018 Mar 30. PMID 29602883